CLINICAL TRIAL: NCT04208581
Title: Yiqi Huoxue Huatan Granule for Reducing Mortality in COPD With Chronic Respiratory Failure: A Randomized, Double-blind, Placebo Controlled Trial
Brief Title: Yiqi Huoxue Huatan Granule for Reducing Mortality in COPD With Chronic Respiratory Failure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking University People's Hospital (Other)
Collaborators: Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Fengcuiling, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM for COPD with CRF
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Respiratory Failure
Keywords: Chronic Obstructive Pulmonary Disease; Chronic Respiratory Failure; Yiqi Huoxue Huatan Granule
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation; Salmeterol Xinafoate; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yiqi Huoxue Huatan granule plus Western medicine (Experimental): Patients in this arm will receive Yiqi Huoxue Huatan granule in addition to Western medicine.
  Interventions: Drug: Yiqi Huoxue Huatan granule
- Placebo Yiqi Huoxue Huatan granule plus Western medicine (Placebo Comparator): Patients in this arm will receive placebo Yiqi Huoxue Huatan granule in addition to Western medicine.
  Interventions: Drug: Placebo Yiqi Huoxue Huatan granule

INTERVENTIONS:
Drug: Yiqi Huoxue Huatan granule — Yiqi Huoxue Huatan granule will be administered twice daily for five days a week for 52 weeks,Tiotropium Bromide Powder for Inhalation will be used once daily (18 μg each time) for 52 weeks, Salmeterol / Fluticasone Powder for Inhalation will be used twice daily (50ug/250ug each time) for 52 weeks, Budesonide / Formoterol Powder for Inhalation will be used twice daily (320ug/4.5ug each time) for 52 weeks.
  Other Names: Tiotropium Bromide Powder for Inhalation; Salmeterol / Fluticasone Powder for Inhalation or Budesonide / Formoterol Powder for Inhalation
  Arms: Yiqi Huoxue Huatan granule plus Western medicine
Drug: Placebo Yiqi Huoxue Huatan granule — Placebo Yiqi Huoxue Huatan granule will be administered twice daily for five days a week for 52 weeks,Tiotropium Bromide Powder for Inhalation will be used once daily (18 μg each time) for 52 weeks, Salmeterol / Fluticasone Powder for Inhalation will be used twice daily (50ug/250ug each time) for 52 weeks, Budesonide / Formoterol Powder for Inhalation will be used twice daily (320ug/4.5ug each time) for 52 weeks.
  Other Names: Tiotropium Bromide Powder for Inhalation; Salmeterol / Fluticasone Powder for Inhalation or Budesonide / Formoterol Powder for Inhalation
  Arms: Placebo Yiqi Huoxue Huatan granule plus Western medicine

SUMMARY:
This study aims to establish the treatment scheme of Yiqi Huoxue Huatan granule for chronic obstructive pulmonary disease (COPD) with chronic respiratory failure (CRF), reducing mortality, improving quality of life and forming high quality evidence.

DETAILED DESCRIPTION:
COPD is a highly prevalent disease, with a prevalence among people 40 years of age or older of 10.1% worldwide and 13.7% in China. COPD has become the third leading cause of death worldwide. COPD complicated by CRF is serious and has a high mortality rate. At present, ideal and effective treatment is inadequate. Traditional Chinese medicine (TCM) has some potential in improving outcomes in COPD with CRF.

This is a multicenter, randomized, double-blind, placebo controlled trial to evaluate the effect of Yiqi Huoxue Huatan granule on reducing mortality and improving quality of life in COPD with CRF. After a 14-day run-in period, 372 subjects will be randomly assigned to treatment group or control group for 52-week treatment, followed by 52-week follow-up. The primary outcomes are all-cause mortality and frequency of acute exacerbation of COPD. The secondary outcomes include clinical symptoms, COPD assessment test (CAT), arterial blood gas analysis, pulmonary function and duration of mechanical ventilation. Safety will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of stable COPD;

  * Arterial blood gas analysis meets criteria of PaO2 < 60mmHg and PaCO2 > 50mmHg during quiet breathing at sea level;
  * Syndrome differentiation meets criteria of Qi deficiency, blood stasis and phlegm turbidity obstructing orifice syndrome；
  * Age ranges from 40 years to 80 years;
  * With informed consent signed.

Exclusion Criteria:

* • CRF resulting from other respiratory diseases, such as bronchiectasis, pulmonary cystic fibrosis, lung cancer, etc.;

  * Acute exacerbation of CRF；
  * Patients with severe cardiovascular and cerebrovascular diseases;
  * Pregnant and lactating women;
  * Patients with psychiatric disorders；
  * Patients with diabetes;
  * Patients who have participated in other clinical studies in the past 4 weeks;
  * Patients who have experienced one or more acute exacerbation of COPD in the past 4 weeks.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Up to week 52 of the follow-up phase.
  All-cause mortality will be calculated in this study.
Frequency of acute exacerbation of COPD | Up to week 52 of the follow-up phase.
  Frequency of acute exacerbation of COPD will be recorded.

SECONDARY OUTCOMES:
Clinical symptom assessment questionnaire | Change from baseline clinical symptom assessment questionnaire scores at week 13, 26, 39 and 52 of the treatment phase, and week 13, 26, 39 and 52 of the follow-up phase.
  Clinical symptom assessment questionnaire of COPD will be used to assess symptoms.
CAT | Change from baseline CAT scores at week 13, 26, 39 and 52 of the treatment phase, and week 13, 26, 39 and 52 of the follow-up phase.
  COPD assessment test (CAT) will be used to assess quality of life.
Arterial partial pressure of oxygen (PaO2) | Change from baseline PaO2 at week 13, 26, 39 and 52 of the treatment phase, and week 13, 26, 39 and 52 of the follow-up phase.
  PaO2 will be evaluated by arterial blood gas analysis.
Arterial partial pressure of carbon dioxide (PaCO2) | Change from baseline PaCO2 at week 13, 26, 39 and 52 of the treatment phase, and week 13, 26, 39 and 52 of the follow-up phase.
  PaCO2 will be evaluated by arterial blood gas analysis.
FEV1 | Change from baseline FEV1 at week 52 of the treatment phase, and week 52 of the follow-up phase.
  Forced expiratory volume in one second ( FEV1) will be used to assess pulmonary function.
Duration of mechanical ventilation | Change from baseline duration of mechanical ventilation at week 13, 26, 39 and 52 of the treatment phase, and week 13, 26, 39 and 52 of the follow-up phase.
  The duration of mechanical ventilation will be recorded.
Health economics | Up to week 52 of the follow-up phase.
  Cost of the treatment phase and follow-up phase will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Suyun Li, Doctor, Study Chair — The First Affiliated Hospital of Henan University of Chinese Medicine
Locations (1):
- Beijing Changping TCM Hospital, Beijing, China

REFERENCES:
- [Derived] Yang JY, Wang HT, Zhao KM, Yu XQ, Huang DH, Wang HX, Wei GS, Bai L, Hou YJ, Huang QT, Hu J, Zhu HZ, Wu L, Lu XC, Chen YF, Gao F, Su LH, Wang Y, Li CY, Li SY, Feng CL. The efficacy and safety of Yiqi Huoxue Huatan granule in the treatment of stable COPD with chronic respiratory failure: A randomized, double-blind, placebo controlled trial. J Ethnopharmacol. 2025 Aug 29;352:120228. doi: 10.1016/j.jep.2025.120228. Epub 2025 Jul 1. PMID 40609812